## Statistical Analysis Plan

Tests of differences will be conducted for comparisons between the INSIGHT Program group and the control group on demographic, penal and outcome variables at baseline. Moreover, tests of differences will also be used to compare the two conditions at postintervention and 3-month follow-up. Within-group differences in outcomes will also be tested. Lastly, Reliable Change Index (RCI; Jacobson & Truax, 1991) will be calculated to measure the intra-subject clinical change. The RCI was created to evaluate the effectiveness of a particular treatment, providing information about treatment effects for each subject. Furthermore, it allows the researcher to understand whether the changes observed in each participant are in fact genuine or just due to measurement errors. The RCI scores will be interpreted based on established criteria: individuals who achieved scores exceeding 0.84 were allocated to the "global improvement" (GI) group, those scoring below -0.84 were placed in the "global deterioration" (GD) group, and those with scores between these values were assigned to the "no change" (NC) category.